CLINICAL TRIAL: NCT02409095
Title: A Phase IV, Non-Inferiority, Observer Blind, Randomized Clinical Study Comparing Safety And Immunogenicity Of DTP-HB-Hib Vaccination by Disposable-Syringe Jet Injector To Vaccination By Needle And Syringe In Healthy Infants In India
Brief Title: Study Comparing DTP-HB-Hib by Disposable-Syringe Jet Injector To Vaccination By Needle And Syringe In Infants
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to increased rate of local injection site reactions in the DSJI group.
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Penta-01/12
Record Dates: First submitted 2015-01-12; First posted 2015-04-06 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Immune Response to DTP-HB-Hib Vaccine
MeSH Terms: interventions — Pentavac; Needles; Syringes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DISPOSABLE-SYRINGE JET INJECTOR (DSJI) (Experimental): Subjects in this arm will be given three deep intramuscular doses, 0.5 mL each dose 4 weeks apart, of Serum Institute of India Ltd.'s DTP-HB-Hib vaccine (Brand name: Pentavac) via Disposable Syringe Jet Injector (Brand Name:Stratis) of Pharmajet Inc
  Interventions: Biological: DTP-HB-Hib vaccine; Device: Disposable Syringe Jet Injector (DSJI)
- NEEDLE & SYRINGE (N-S) (Active Comparator): Subjects in this arm will be given three deep intramuscular doses, 0.5 mL each dose 4 weeks apart, of Serum Institute of India Ltd.'s DTP-HB-Hib vaccine (Brand name: Pentavac) via conventional needle and Syringe
  Interventions: Biological: DTP-HB-Hib vaccine; Other: Needle & Syringe

INTERVENTIONS:
Biological: DTP-HB-Hib vaccine — Diphtheria, Tetanus, Pertussis, Hepatitis-B and Haemophilus influenzae type-B conjugate vaccine (DTP-HB-Hib) has been developed and manufactured by SIIL. The vaccine is pre-qualified by WHO and licensed by the Indian regulatory authority for immunization in children to protect them against above five diseases.
  Other Names: Pentavac
Device: Disposable Syringe Jet Injector (DSJI) — Stratis is a needle free injection device manufactured by Pharamjet Inc. and licensed in USA.
  Other Names: Stratis
  Arms: DISPOSABLE-SYRINGE JET INJECTOR (DSJI)
Other: Needle & Syringe — The conventional needle syringe that is routinely used for vaccination.
  Arms: NEEDLE & SYRINGE (N-S)

SUMMARY:
This is a study planned to determine and compare immunogenicity and reactogenicity of DTP-HB-Hib vaccine of SIIL delivered either with disposable-Syringe Jet Injector (DSJI) or disposable-syringe needle in total 340 Indian infants aged 6 to 8 weeks at the time of enrollment.

It will provide information to aid managers, device regulatory control officials, immunization programs, and clinicians who make decisions on safe clinical practice standards.

DETAILED DESCRIPTION:
This is a randomized, observer blind, non-inferior, parallel group, multi-centre clinical study to determine and compare immunogenicity and reactogenicity of DTP-HB-Hib vaccine of Serum Institute of India Ltd. delivered either with disposable-Syringe Jet Injector (DSJI) or disposable-syringe needle in total 340 Indian infants. Sera samples will be analyzed by ELISA for seroconversion / seropositivity for each individual component of vaccine i.e. Diphtheria, Tetanus, Pertussis, Hepatitis B (HBsAg) and Hemophilus Influenza B at 28 days after administration of a third dose of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy infants of age 6-8 weeks at the time of the first vaccination.
2. Born after a normal gestation period (36-42 weeks).
3. Parents of subjects willing to give written informed consent.
4. Parents willing to comply with study protocol.
5. Free of obvious health problems as established by medical history and screening evaluation including clinical examination.
6. The participant should be the resident of study area

Exclusion Criteria:

1. Infant subject participating in other clinical trial or planned participation in another clinical trial during the present trial period.
2. Infant with congenital or acquired immunodeficiency, malignancy or receiving immunosuppressive therapy such as systemic corticosteroids therapy for a period of ≥ 1 week.
3. Infant with history of allergy or systemic hypersensitivity to any of the vaccine component or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
4. Infant with any chronic illness including hepatic, renal, respiratory, CVS, endocrine and neurological illness.
5. Infants who have received blood or blood-derived products in the past.
6. History of diphtheria, tetanus, pertussis, and hepatitis B or Haemophilus influenzae type b (confirmed either clinically, serologically or microbiologically).
7. Previous history of vaccination against the diphtheria, tetanus, pertussis or Hib.
8. Known history of a bleeding disorder contraindicating intramuscular vaccination.
9. History of any neurological disorder or history of seizure (febrile or afebrile), or encephalopathy, encephalitis, hypotonic-hyporesponsive episode.
10. History of febrile illness at the time of inclusion is a temporary exclusion criterion.
11. Acute or chronic, clinically significant pulmonary, endocrine, autoimmune, cardiovascular, metabolic, hepatic or renal functional abnormality, as determined by medical history, and physical examination tests, which in the opinion of the investigator, might interfere with the study objectives
12. Infant with any other condition, which, in the opinion of the investigator would jeopardize the safety or rights of the infant participating in the study or making it unlikely the subject could complete the protocol

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of seroprotection and geometric mean titers (GMT) for diphtheria, tetanus, hepatitis-B, H. Influenzae and percentage sero-positivity and GMT for B. Pertussis | one month after administration of third dose of the vaccine

SECONDARY OUTCOMES:
Occurrence of solicited reactions | within 4 days following the administration of each of the three vaccine dose
Occurrence of adverse event | 84 days after first vccine dose
Occurrence of serious adverse event | 84 days after first vccine dose

CONTACTS AND LOCATIONS:
Locations (3):
- India (3):
  - Department of Pediatrics, KEM Hospital Research Centre, Sardar Moodliar Road, Rasta Peth,, Pune, Maharashtr
  - Department of Pediatrics, Bharati Vidyapeeth Deemed University Medical College and Hospital, Satara Road, Katraj, Dhankawadi, Pune, Maharasthra
  - Dept of Pediatrics, Sri Ramachandra Medical Centre, No. 1, Ramachandra nagar, Porur,, Chennai, Tamil Nadu

REFERENCES:
- [Derived] Bavdekar A, Malshe N, Ravichandran L, Sapru A, Kawade A, Lalwani S, Palkar S, Hanumante N, Gunale B, Kapse D, Chaudhari A, Miller T, Saganic L, Jarrahian C, McGray S, Zehrung D, Kulkarni PS. Clinical study of safety and immunogenicity of pentavalent DTP-HB-Hib vaccine administered by disposable-syringe jet injector in India. Contemp Clin Trials Commun. 2019 Jan 9;14:100321. doi: 10.1016/j.conctc.2019.100321. eCollection 2019 Jun. PMID 30899835